CLINICAL TRIAL: NCT00819572
Title: A Double-blind, Randomised, Placebo-controlled Phase I/IIa Study to Investigate the Safety, Tolerability and Efficacy on Pain of Intra-articular DLX105 Applied to Patients With Severely Painful Osteoarthritis of the Knee
Brief Title: Study of Intra-articular DLX105 Applied to Patients With Severely Painful Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ESBATech AG (Industry)
Responsible Party: Hamish Cameron, CEO, Delenex AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLX105CRD02
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; TNF-alpha; DLX105; scFv antibody fragment; pain; fragment; antibody fragment
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): DLX105 low dose
  Interventions: Biological: DLX105, a single-chain (scFv) antibody fragment against TNF-alpha
- 2 (Experimental): DLX105 high dose
  Interventions: Biological: DLX105, a single-chain (scFv) antibody fragment against TNF-alpha
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: DLX105, a single-chain (scFv) antibody fragment against TNF-alpha — Comparison of two different doses of intra-articular DLX105
  Arms: 1; 2
Drug: Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether an intra-articular injection of DLX105 to the knee joint of patients suffering from severly painful osteoarthritis is safe and reduces pain.

DETAILED DESCRIPTION:
Treatment options for patients suffering from osteoarthritis remain limited. TNF-alpha has been identified as a major pro-inflammatory component inducing and perpetuating peripheral hyperalgesia and cartilage degeneration in various preclinical studies. DLX105 is an antibody fragment of comparably low molecular weight, associated with an exceptional local biodistribution pattern upon intra-articular injection. In addition, due to its short systemic half life as compared to conventional monoclonal antibodies, systemic exposure to DLX105 upon intra-articular administration is low. This study is designed to determine the safety and local tolerability profile of single intra-articular injections of ESBA105 as well as to define DLX105's effect size and effect duration in reducing pain of patients suffering from severely painful osteoarthritis of the knee. The study will be conducted in two sequential parts. In a first part, 4 different doses of DLX105 will be compared in a sequential, escalating scheme against placebo treatment in a total of 24 patients. In the second part of the study, two doses of DLX105 chosen based on safety data from the first part will be compared to placebo treatment in a total of 102 patients.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 30.
* Patients with diagnosed OA of the knee (unilateral or bilateral) according to the American College of Rheumatology (ACR) Criteria for classification of idiopathic OA (clinical and radiological criteria) of the knee at Screening (for ACR criteria, see Appendix 16.1).
* Radiographic evidence of tibiofemoral OA within the last 6 months before Screening, consisting of Grade II or Grade III changes, according to Kellgren-Lawrence grading system.
* Presence of pain in the index knee (in case of bilateral OA, "index knee" is the more painful knee) defined by a level of ≥ 60 mm on a 100 mm (linear) VAS at Screening.
* Paracetamol and NSAIDs (apart from acetyl salicylic acid ≤ 100 mg/day) must be withdrawn at least 24 hours prior to Screening .
* Doses of "chondroprotective" agents containing glucosamine and/or chondroitin sulphate must be stable for at least 3 months prior to Screening.
* Doses of any non-prescription medication claiming effects on signs or symptoms of OA must be stable for at least 3 months prior to Screening.
* Use of non-pharmacological treatment modalities must be stable for at least 3 months prior to Screening.
* Negative QuantiFERON-TB Gold test.

Exclusion Criteria:

* Radiographic evidence of tibiofemoral OA within the last 6 months before Screening, consisting of Grade IV, according to Kellgren-Lawrence grading system.
* Instability of the index knee joint of > 10° as assessed by goniometer at Screening.
* Arthroscopic or open surgery to the index knee joint within 6 months prior to Screening.
* Post-traumatic or any other secondary OA of the knee.
* Isolated OA of the patello-femoral joint.
* Co-morbidity that would confound measurement of knee pain
* Evidence of any inflammatory arthritis.
* History of Reiter's Syndrome, RA, psoriatic arthritis, ankylosing spondylitis, lymphoma, arthritis associated with inflammatory bowel disease, sarcoidosis, amyloidosis, or any other inflammatory disease (immune mediated inflammatory disease) that may affect the knee.
* Local or systemic contraindication for an i.a. injection at Screening or Baseline.
* Any i.a. injection (corticosteroids, hyaluronic acid, etc.) within the 3 months prior to Screening.
* History of high risk exposure to Mycobacterium tuberculosis.
* Human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection.
* Uncontrolled diabetes or cardiovascular disease (New York Heart Association criteria III + IV), including uncontrolled hypertension (> 160/100 mmHg).
* Active infectious episodes, or history of recurrent or chronic systemic infections.
* Malignancy within 5 years prior to Screening, except for surgically-cured non melanoma skin cancer or cervical carcinoma in situ.
* Significant haematological disease within 1 month prior to Screening.
* Moderately to severely impaired hepatic function, or laboratory values reflecting inadequate hepatic function

Additional criteria for the sub-population of patients undergoing MRI:

* Contraindications to MRI.
* Known allergy to gadolinium contrast material.
* Presence of chronic renal failure defined by a calculated creatinine clearance (CrCl) of < 60 mL/min, using the Cockcroft-Gault estimate for GFR

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (Day 0) to Day 7 in a 100mm Visual Analogue Scale (VAS) to assess the intensity of knee pain. | Day 7 after intra-articular injection
Safety assessment during the study period. Safety endpoints will include the nature and incidence of AEs, physical examination findings, changes in vital signs, and laboratory test results. | 8 weeks / 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis (WOMAC™) scoring | Day 7 after intra-articular injection

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Georg Schett, MD, Study Chair — University Hospital of Erlangen, Germany; Prof. Hansjörg Häuselmann, MD, Principal Investigator — Rheumazentrum, Zurich Switzerland (Country Coordinator); PD.Dr. Diego Kyburz, MD, Principal Investigator — University Hospital Zurich, Switzerland (Country Coordinator)
Locations (10):
- Germany (4):
  - Prof. Dr. med. Georg Schett, Erlangen
  - Dr. René Martz, Hamburg
  - Dr. Sven Ostermeier, Hanover
  - Prof. Dr. Manfred Hartard, Munich
- Switzerland (6):
  - Rheumaklinik Kantonsspital Aarau, Aarau
  - Rheumatologische Universitäts-Poliklinik, Felix-Platter Spital Basel, Basel
  - Service de rhumatologie, Centre Hospitalier Universitaire, Lausanne, Lausanne
  - Kantonsspital St.Gallen, Rheumatologie, Sankt Gallen
  - Zentrum für Rheuma und Knochenerkrankungen, Zurich
  - Universitätsspital Zürich, Rheumaklinik, Zurich